CLINICAL TRIAL: NCT04242563
Title: Virtual Reality for Preoperative Anxiety in Interventional Cardiology
Acronym: No PANIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC19.116
Record Dates: First submitted 2019-12-30; First posted 2020-01-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: interventional cardiopathy; preoperative anxiety; virtual reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): No virtual reality
- INTERVENTION GROUP (Experimental): Patient equipped with Virtual reality in transfer room.
  Interventions: Other: VIRTUAL REALITY

INTERVENTIONS:
Other: VIRTUAL REALITY — Patient equipped with virtual reality in transfer room
  Arms: INTERVENTION GROUP

SUMMARY:
Improving the management of perioperative anxiety is important. Anxiety can have an impact on the intervention and can increase postoperative complications as well as emotional and behavioral incidents that then have an impact on adherence to care. These findings are also true in interventional cardiology. That is why, for several months, the Grenoble University hospital paramedical team, in collaboration with the medical profession, improved by using several techniques (educational sheet, therapeutic communication). Following a survey of the patients of Grenoble university hospital, a gray area persists in their care. The room where the patient attends his examination. The investigators would then use the new technology that makes virtual reality in the transfer room to evaluate its benefit in a random study on preoperative anxiety in interventional cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Major male or female patient
* Coronarography procedure programmed for exploration of coronary artery disease following a positive ischemia test, realized in ambulatory
* Patient who has given written consent to participate in the study

Exclusion Criteria:

* Arrhythmia patient and / or patient with a pacemaker
* Hemodynamic instability
* Patient who has already had coronarography
* Prior revascularization by coronary bypass
* End-stage renal disease (Creatinine clearance <30 ml / min),
* Allergy to iodine contrast agent
* Blind or visually impaired patient (high degree)
* Deaf or hard of hearing patient
* Patient with claustrophobia or unable to wear a mask over the eyes
* Patient whose physical or psychological state could compromise obtaining informed consent and compliance with protocol requirements
* Patient under administrative or judicial supervision
* Foreign patient who does not understand French
* Major patient protected by law (article L1121-8 and L1121-5)
* Pregnant or lactating patient
* Patient not affiliated with social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of virutal reality on the management of preoperative anxiety measured by heart rate variability in interventional cardiology room in patient awaiting coronarography | Time 1 : 60 minutes
  Heart rate variability during 20 minutes by a heart rate monitor in transfer room

SECONDARY OUTCOMES:
Evaluation of anxiety level in patient awaiting coronarography | TIme 1 : 60 minutes, Time 2 : 120 minutes
  The Analogical Self-Assessment Scale for Preoperative Anxiety (0 - no anxiety to 10 - uncontrollable anxiety)
Patient satisfaction on the global care in the coronary angiography room | Time 3 : 180 minutes
  Patient satisfaction questionnaire
Impact of virtual reality on coronarography intervention duration | Time 2 : 120 minutes
  Intervention duration (in minutes)
Impact of virtual reality on coronarography irradiation dose | Time 2 : 120 minutes
  Irradiation dose (in Gy.cm²)
Impact of virtual reality on coronarography scopy time | Time 2 : 120 minutes
  scopy time (in minutes)
Impact of virtual reality on administration of analgesic and anxiolytic drug peri and per coronarography procedure | Time 2 : 120 minutes
  administration of analgesic and anxiolytic drug peri and perprocedure (drug name and dose)
Impact of virtual reality on rate and success of coronarography procedure | Time 2 : 120 minutes
  number and success of PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Larsson CE, Cabassut V, Peretout P, Marliere S, Vautrin E, Piliero N, Salvat M, Riou L, Vanzetto G, Vilotitch A, Bosson JL, Barone-Rochette G. Assessment of the Objective Effect of Virtual Reality for Preoperative Anxiety in Interventional Cardiology. Am J Cardiol. 2023 Oct 15;205:207-213. doi: 10.1016/j.amjcard.2023.07.130. Epub 2023 Aug 21. PMID 37611412